CLINICAL TRIAL: NCT03574831
Title: the Efficency and Safety of the Endoscopic Radiofrequency Procedure in Gastroesophageal Reflux Diseases
Brief Title: the Efficency and Safety of Stretta in GERD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Guo Zihao, Clinical Professor, Capital Medical University
Other Study IDs: xhnk001
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: GERD; Radiofrequency Ablation
Keywords: GERD; Radiofrequency ablation; efficiency; safety
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stretta: Radio Frequency Ablation (RFA) using a Stretta device.
  Interventions: Device: Stretta

INTERVENTIONS:
Device: Stretta — Stretta

SUMMARY:
This study evaluated the efficency and safety of the endoscopic radiofrequency procedure(Stretta) in adult gastroesophageal patients.

DETAILED DESCRIPTION:
Gastro-esophageal reflux disease (GERD) is the most common outpatient diagnosis in gastroenterology and is associated with a significant burden on the healthcare system. Proton pump inhibitors (PPIs) are the mainstay of GERD treatment,howerver, some patients have an unsatisfactory response to high doses of PPIs, which remains a challenge. The Stretta procedure, a radiofrequency (RF) application to the lower esophageal sphincter (LES), was introduced about 15 years ago as an alternative to chronic medical therapy or surgical intervention for GERD.The Stretta procedure appears to result in thickening of the LES, decreased transient LES relaxation rate and reduced esophageal acid exposure.The majority studies of Stretta were held in USA and Europe, the sduty of Stretta in Asia is rare. The investigators propose to perform a prospectively observiton study to evaluate the efficency of the Stretta procedure in patients of refractory GERD in China.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Small hiatus hernia (< 2-3 cm)
3. Los Angeles Grade 'A' or 'B' Reflux Esophagitis or non erosive esophagitis
4. LES pressure <15 mm Hg
5. PPI dependent / refractory GERD
6. abnormal 24h esophagus pH-impedance monitoring

Exclusion Criteria:

1. Age < 18 years
2. Large hiatus hernia (> 3 cm)
3. Los Angeles Grade 'C' or 'D' Reflux Esophagitis
4. LES pressure > 15 mm Hg
5. Underlying coagulation disorder
6. Previous Esophageal or Gastric surgery
7. Pregnant
8. major esophagus motility disorder according to Chicago v3.0

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with refractory GERD symptoms, without major esophagus motility disorder and large hiatus hernia.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-01-02 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
GERD-HRQL scores | [Time Frame: Change from Baseline HRQL scores at 1 month;Change from Baseline HRQL scores at 2 months;Change from Baseline HRQL scores at 6 months;Change from Baseline HRQL scores at 1 year]
  the improvement of GERD-HRQL scores after procedure.Scale ranges 0-50 points, the lower score means the better efficacy.

SECONDARY OUTCOMES:
Number of patients who report independence from Proton Pump Inhibitor (PPI) drug post Stretta procedure | Change from Baseline number at 1 month;Change from Baseline number at 2 months;Change from Baseline number at 6 months;Change from Baseline number at 1 year]
  Questionnaire will be provided to each participant to report no further requirement of PPI drug post procedure.
Demeester Score | 1 year
  the change of Demeester scores after procedure. The lower, the better.
LES Pressure | 1 year
  the change of LES pressure after procedure.The higher, the better.
Number of participants with treatment-related adverse events | 1 month
  Number of participants with treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Chuan Zhang, MD, Study Chair — Gatroenterology department,Beijing Tong Ren Hospital, Capital Medical University
Locations (1):
- Gastroenterology department,Beijing Tong Ren Hospital, Capital Medical University., Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided